CLINICAL TRIAL: NCT00615433
Title: A Phase 3 Randomized, Placebo-and Active Comparator Controlled, Clinical Trial to Study the Safety and Efficacy of Two Doses of Lurasidone HCl in Acutely Psychotic Patients With Schizophrenia.
Brief Title: Lurasidone HCl A Phase 3 Study of Patients With Acute Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D1050231
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Results first posted 2011-02-14 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-05

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Latuda; Lurasidone
MeSH Terms: conditions — Schizophrenia | interventions — Lurasidone Hydrochloride; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Lurasdione 40mg tablets (Experimental)
  Interventions: Drug: Lurasidone 40 mg tablets
- 120mg (Experimental)
  Interventions: Drug: Lurasidone
- 15mg Olz (Active Comparator)
  Interventions: Drug: Olanzapine
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: Lurasidone — 120mg/day
  Arms: 120mg
Drug: Olanzapine — 15mg/day
  Arms: 15mg Olz
Drug: Placebo comparator — Placebor Comparator
  Arms: Sugar pill
Drug: Lurasidone 40 mg tablets — Lurasidone 40 mg tablets
  Arms: Lurasdione 40mg tablets

SUMMARY:
Lurasidone HCl is a compound developed for the treatment of schizophrenia. This clinical study is designed to test the hypothesis that lurasidone is more efficacious than placebo. The study will also evaluate the safety and tolerability of lurasidone as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent and aged between 18 and 75 years of age.
* Meets DSM-IV criteria for a primary diagnosis of schizophrenia.
* Not pregnant, if of reproductive potential agrees to remain abstinent or use adequate and reliable contraception for duration of study.
* Able and agrees to remain off prior antipsychotic medication for the duration of study.
* Good physical health on the basis of medical history, physical examination, and laboratory screening.
* Willing and able to comply with the protocol, including the inpatient requirements and outpatient visits.

Exclusion Criteria:

* Considered by the investigator to be at imminent risk of suicide or injury to self, others or property.
* Any chronic organic disease of the CNS (other than schizophrenia).
* Used investigational compound within 30 days.
* Clinically significant or history of alcohol abuse/alcoholism or drug abuse/dependence within the last 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Actual)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (52):
- United States (25):
  - K&S Professional Research Services LLC, Little Rock, Arkansas
  - Woodland International Research Group, LLC, Little Rock, Arkansas
  - Clinical Pharmacological Studies, Inc., Cerritos, California
  - Excell Research, Oceanside, California
  - University of California at Irvine Medical Center, Orange, California
  - California Clinical Trials, Paramount, California
  - CNRI - San Diego, LLC, San Diego, California
  - UCSD Medical Center, San Diego, California
  - Collaborative Neuroscience Network Inc., Torrance, California
  - Florida Clinical Research Center, LLC, Fruitland Park, Florida
  - Segal Institute for Clinical Research, North Miami, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Uptown Research Institute, LLC, Chicago, Illinois
  - Alexian Brothers Health System, Hoffman Estates, Illinois
  - Lousiana Clinical Research, LLC, Shreveport, Louisiana
  - Precise Research Center, Flowood, Mississippi
  - St. Charles Psychiatric Associates-Midwest Research, Saint Charles, Missouri
  - St. Louis Clinical Trials, St Louis, Missouri
  - CRI Worldwide @ Lourdes, Willingboro, New Jersey
  - Neurobehavioral Research Inc., Cedarhurst, New York
  - University of North Carolina at Chapel Hill, Raleigh, North Carolina
  - Keystone Clinical Studies, LLC, Norristown, Pennsylvania
  - Vanderbilt Heart and Vascular Institute, Nashville, Tennessee
  - Community Clinical Research, Inc., Austin, Texas
  - Claghorn-Lesem Research Clinic, Inc., Houston, Texas
- Colombia (5):
  - Instituto Colombiano del Sistema Nervioso Clinica Montserrat, Cundinamarca, Bogota D.C.
  - CIPNA Centro de Investigaciones y Proyectos en Neurociencias, Barranquilla
  - Centro de Investigacion y Atencion para la Salud Mental, Bogotá
  - Centro de Investigaciones del Sistema Nervioso Limitada, Bogotá
  - Psynapsis Salud Mental, S.A., Risaralda
- India (14):
  - Vijayawada Institute of Mental Health and Neurosciences, Vijaywada, Andh Prad
  - Government Hospital for Mental Care, Visakhapatnam, Andh Prad
  - Hospital for Mental Health - Dept of Psychiatry, Ahmedabad, Gujarat
  - Sheth Vadilal Sarabhai General Hospital, Ahmedabad, Gujarat
  - SBKS Medical College and Brij Psychiatry Hospital, Vadodara, Gujarat
  - Victoria Hospital, Bangalore, Karna
  - Kasturba Medical College, Mangalore, Karna
  - Father Muller Institute of Medical Education and Research, Mangalore, Karna
  - Justice K.S. Hedge Charitable Hospital, Mangalore, Karna
  - Kasturba Hospital, Manipal, Karna
  - JSS Medical College and Hospital - Dept of Psychiatry, Mysore, Karna
  - Shanti Nursing Home, Aurangabad, Mahara
  - Deenanath Mangeshkar Hospital, Pune, Mahara
  - Madras Medical College & Government General Hospital, Chennai, Tamil Nadu
- Lithuania (4):
  - Ziegzdriai Mental Hospital, Public Institution, Kaunas
  - Klaipeda Mental Hospital, Public Institution, Klaipėda
  - Siauliai Mental Hospital, Public Institution, Šiauliai
  - Republican Vilnius Psychiatry Hospital, Public Institution, Vilnius
- Philippines (4):
  - Davao Medical School Foundation Hospital, Davao City
  - Makati Medical Center, Makati City
  - National Center for Mental Health, Mandaluyong
  - Metro Psych Facility, Mandaue City

REFERENCES:
- [Background] Meltzer HY, Cucchiaro J, Silva R, Ogasa M, Phillips D, Xu J, Kalali AH, Schweizer E, Pikalov A, Loebel A. Lurasidone in the treatment of schizophrenia: a randomized, double-blind, placebo- and olanzapine-controlled study. Am J Psychiatry. 2011 Sep;168(9):957-67. doi: 10.1176/appi.ajp.2011.10060907. Epub 2011 Jun 15. PMID 21676992
- [Result] Stahl SM, Cucchiaro J, Simonelli D, Hsu J, Pikalov A, Loebel A. Effectiveness of lurasidone for patients with schizophrenia following 6 weeks of acute treatment with lurasidone, olanzapine, or placebo: a 6-month, open-label, extension study. J Clin Psychiatry. 2013 May;74(5):507-15. doi: 10.4088/JCP.12m08084. Epub 2013 Mar 13. PMID 23541189
- [Derived] Hopkins SC, Tomioka S, Ogirala A, Loebel A, Koblan KS, Marder SR. Assessment of Negative Symptoms in Clinical Trials of Acute Schizophrenia: Test of a Novel Enrichment Strategy. Schizophr Bull Open. 2022 Apr 7;3(1):sgac027. doi: 10.1093/schizbullopen/sgac027. eCollection 2022 Jan. PMID 39144777
- [Derived] Hopkins SC, Ogirala A, Worden M, Koblan KS. Depicting Safety Profile of TAAR1 Agonist Ulotaront Relative to Reactions Anticipated for a Dopamine D2-Based Pharmacological Class in FAERS. Clin Drug Investig. 2021 Dec;41(12):1067-1073. doi: 10.1007/s40261-021-01094-7. Epub 2021 Nov 9. PMID 34751928
- [Derived] Nasrallah HA, Cucchiaro JB, Mao Y, Pikalov AA, Loebel AD. Lurasidone for the treatment of depressive symptoms in schizophrenia: analysis of 4 pooled, 6-week, placebo-controlled studies. CNS Spectr. 2015 Apr;20(2):140-7. doi: 10.1017/S1092852914000285. Epub 2014 Jun 23. PMID 24955752

RESULTS

PARTICIPANT FLOW:
Groups:
- 40mg: Lurasidone 40 mg tablet taken orally once a day. The number of subjects in the participant flow (overall study) is based on the total number of subjects randomized (478). The number of subjects in the baseline characteristics is based on the safety population (475). All randomized subjects who received at least one dose of study medication were included in the safety analysis. One subject who was randomized to the 40 mg treatment group did not take any study medication.
- 120mg: 3 40 mg tablets taken orally once a day. The number of subjects in the participant flow (overall study) is based on the total number of subjects randomized (478). The number of subjects in the baseline characteristics is based on the safety population (475). All randomized subjects who received at least one dose of study medication were included in the safety analysis. One subject who was randomized to the 120 mg treatment group did not take any study medication.
- 15mg Olz: 3 5 mg Olanzapine over-encapsulated capsules taken orally once a day. The number of subjects in the participant flow (overall study) is based on the total number of subjects randomized (478). The number of subjects in the baseline characteristics is based on the safety population (475). All randomized subjects who received at least one dose of study medication were included in the safety analysis. One subject who was randomized to the 15 mg Olanzapine treatment group did not take any study medication.
- Placebo: Placebo to match lurasidone 40mg (tablets or placebo to match olanzapine 5 mg (over-encapsulated).
Period: Overall Study
Arm/Group | 40mg | 120mg | 15mg Olz | Placebo
Started | 120 | 119 | 123 | 116
Completed | 77 | 66 | 84 | 71
Not Completed | 43 | 53 | 39 | 45

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 40mg | 120mg | 15mg Olz | Placebo | Total
Number analyzed (Participants) | 119 | 118 | 122 | 116 | 475
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (11.0) | 37.9 (11.2) | 38.3 (10.2) | 36.9 (11.3) | 37.7 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 27 | 26 | 104
  Male | 93 | 93 | 95 | 90 | 371
Region of Enrollment [Number; unit: participants]
  United States | 70 | 72 | 74 | 68 | 284
  Philippines | 7 | 6 | 8 | 5 | 26
  Lithuania | 7 | 7 | 7 | 8 | 29
  Colombia | 12 | 12 | 12 | 12 | 48
  India | 23 | 21 | 21 | 23 | 88

OUTCOME MEASURES:

1. Primary Outcome: Change in Total PANSS (Positive and Negative Syndrome Scale)Score From Baseline to the End of the Double Blind Treatment Period.
Description: The PANSS is a 30-item rating instrument evaluating the presence/absence and severity of positive, negative and general psychopathology of schizophrenia. The scale was developed from the BPRS and the Psychopathology Rating Scale. All 30 items are rated on a 7-point scale (1=absent; 7=extreme). The total score can range from 30 to 210. Lower scores represent less severity of illness.
Time Frame: Baseline and 6 weeks
Population: The primary population for the efficacy analysis was the Intent-to-Treat (ITT) population. All subjects who were randomized, received at least one dose of study medication, and have a Baseline efficacy measurement and at least one post-Baseline efficacy measurement, were in the efficacy analysis in the treatment group to which they were randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Groups:
- 120mg: 3 40 mg tablets taken orally once a day.
Arm/Group | 40mg | 120mg | 15mg Olz | Placebo
Number analyzed (Participants) | 118 | 118 | 121 | 114
Units on a scale | -25.7 [-29.6 to -21.8] | -23.6 [-27.8 to -19.4] | -28.7 [-32.4 to -24.9] | -16.0 [-20.1 to -12.0]
Statistical Analysis 1: Comparison: 40mg vs 120mg vs Placebo; Improvements in PANSS ratings are estimated from 2 prior studies of lurasidone. Assuming lurasidone differs from placebo in change from baseline in PANSS by 6.8 and 10.0 for 40 and 120 mg, respectively, and assuming a standard deviation of 19.1, then n=120 subjects per group provides approximately 97% power (at α=0.05, two-sided) to reject the null hypothesis of no difference from placebo for at least 1 dose. This calculation uses Bonferroni's procedure for controlling pairwise differences; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis

2. Secondary Outcome: CGI-S (Clinical Global Impression - Severity) Change From Baseline to the End of the Double-blind Treatment.
Description: The CGI-S is a clinician-rated assessment of the subject's current illness state on a 7-point scale, where a higher score is associated with greater illness severity.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: scale
Arm/Group | 40mg | 120mg | 15mg Olz | Placebo
Number analyzed (Participants) | 119 | 118 | 122 | 114
scale | -1.5 [-1.7 to -1.3] | -1.4 [-1.6 to -1.2] | -1.5 [-1.7 to -1.4] | -1.1 [-1.3 to -0.9]
Statistical Analysis 1: Comparison: 40mg vs 120mg vs Placebo; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis

ADVERSE EVENTS:
Arm/Group | 40mg | 120mg | 15mg Olz | Placebo
Serious Adverse Events (participants affected / at risk) | 2/119 | 6/118 | 5/122 | 5/116
Other Adverse Events (participants affected / at risk) | 90/119 | 96/118 | 98/122 | 84/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 40mg (N=119) | 120mg (N=118) | 15mg Olz (N=122) | Placebo (N=116)
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Angina Pectoris (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Heamatemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 1
Panic Attack (Psychiatric disorders) | 0 | 0 | 0 | 1
Psychotic Disorder (Psychiatric disorders) | 0 | 4 | 1 | 1
Schizophrenia (Psychiatric disorders) | 1 | 2 | 1 | 0
Substance Abuse (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 1 | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 40mg (N=119) | 120mg (N=118) | 15mg Olz (N=122) | Placebo (N=116)
Constipation (Gastrointestinal disorders) | 6 | 9 | 8 | 6
Dry Mouth (Gastrointestinal disorders) | 2 | 3 | 12 | 1
Dyspepsia (Gastrointestinal disorders) | 9 | 9 | 5 | 7
Nausea (Gastrointestinal disorders) | 13 | 9 | 6 | 5
Salivary Hypersecretion (Gastrointestinal disorders) | 2 | 8 | 1 | 0
Tootache (Gastrointestinal disorders) | 4 | 3 | 12 | 6
Vomiting (Gastrointestinal disorders) | 5 | 10 | 2 | 8
Weight Increased (Investigations) | 2 | 2 | 25 | 6
Decreased Appetite (Metabolism and nutrition disorders) | 6 | 1 | 2 | 2
Increased Appetite (Metabolism and nutrition disorders) | 1 | 3 | 7 | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 6 | 6 | 7 | 4
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 3 | 6 | 3 | 2
Akathisia (Nervous system disorders) | 14 | 27 | 9 | 1
Dizziness (Nervous system disorders) | 5 | 6 | 3 | 2
Dystonia (Nervous system disorders) | 4 | 9 | 1 | 1
Headache (Nervous system disorders) | 26 | 21 | 17 | 25
Parkinsonism (Nervous system disorders) | 11 | 13 | 6 | 2
Sedation (Nervous system disorders) | 11 | 16 | 17 | 4
Somnolence (Nervous system disorders) | 11 | 18 | 11 | 5
Tremor (Nervous system disorders) | 2 | 9 | 7 | 5
Agitation (Psychiatric disorders) | 13 | 7 | 8 | 6
Anxiety (Psychiatric disorders) | 12 | 12 | 7 | 8
Insomnia (Psychiatric disorders) | 15 | 14 | 13 | 13
Psychotic Disorder (Psychiatric disorders) | 2 | 0 | 3 | 7
Restlessness (Psychiatric disorders) | 6 | 4 | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For multi-center studies, it is mandatory that the first publication is based on all data obtained from all analyses as stipulated in the protocol. Investigators participating in multicenter studies must agree not to present data gathered individually or by subgroup of centers before the full, initial publication, unless this has been agreed to by all other investigators and also by Sunovion.